CLINICAL TRIAL: NCT04647240
Title: A Two Part, Randomized Study of Dermacyte® Amniotic Wound Care Liquid for the Treatment of Non-Healing Venous Stasis Ulcers
Brief Title: Dermacyte® Amniotic Wound Care Liquid for the Treatment of Non-Healing Venous Stasis Ulcers
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Merakris Therapeutics (Industry)
Collaborators: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DL-VSU-201
Record Dates: First submitted 2020-11-22; First posted 2020-11-30 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Venous Stasis Ulcer; Venous Leg Ulcer
MeSH Terms: conditions — Varicose Ulcer

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dermacyte® Liquid (human amniotic fluid) (Active Comparator): Dermacyte® Liquid (human amniotic fluid) solution 1.0mL to 2.0mL weekly
  Interventions: Biological: Dermacyte® Liquid (human amniotic fluid)
- Placebo (0.9% saline) (Placebo Comparator): Matching placebo solution 1.0mL to 2.0mL weekly
  Interventions: Biological: Dermacyte® Liquid (human amniotic fluid)

INTERVENTIONS:
Biological: Dermacyte® Liquid (human amniotic fluid) — Subcutaneous injection into and/or around wound bed weekly

SUMMARY:
DL-VSU-201 is a randomized, double-blind, placebo controlled study in subjects with a non-infected venous stasis ulcer (VSU) that has failed to demonstrate improvement after receiving at least 4 weeks of standard, conventional wound therapy to evaluate the efficacy and safety of Dermacyte® Liquid (MTX-001).

DETAILED DESCRIPTION:
DL-VSU-201 is a multi-center, two-part study in patients with VSU (n=40). The run-in phase of the study (Part 1) will enroll 10 eligible subjects. In part 1, patients will be randomized 1:1 to receive active Dermacyte once weekly or once every two weeks with standard of care. The data from Part 1 will be reviewed to determine the administration frequency of the study product (once weekly or once every two weeks) in Part 2 of the Study.

In Part 2, approximately 30 subjects will be randomized 1:1 to receive Dermacyte Liquid or placebo (0.9% NaCl) with standard of care. Subjects will be followed for 12 weeks.

Subjects will receive localized subcutaneous injection of Dermacyte® Liquid or placebo into and/or around the wound bed during during clinic visits over a 12-week period and assessed for safety and efficacy measures at Screening, Baseline, and Weeks 4, 8, and 12. Percent reduction of the wound surface area will be formally collected at Baseline, Weeks 4, 8, and 12. To assess healing, the ulcer will be evaluated by assessing the change in the surface area (L X W) from Baseline. Overall change in VAS from Baseline to Week 12 will be evaluated and total wound closure will be evaluated at Week 12.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who voluntary give written informed consent to participate in study
* Males and female subjects aged 18 to 75 years inclusive at Screening (date the subject provides written informed consent to participate in study) for Part 1 only
* Males and female subjects aged 18 to 80 years inclusive at Screening (date the subject provides written informed consent to participate in study) for Part 2 only
* Subjects must have a full thickness ulcer that meets the following criteria:

  * Ulcer surface area > 1 cm2 and < 25 cm2
  * Ulcer surface area hasn't increased or decreased by 25% or more, as assessed within 14 days or more prior to Baseline
  * Ulcer depth > 0.2 cm at the deepest point of the wound, as measured by gently inserting a pre-moistened cotton tipped applicator into the deepest part of the wound.
  * Ulcer age < 12 months (365 days) prior to Baseline (for Part 2 only)
* Received > 28 days of standard, conventional wound therapy with a high-compression, multilayer bandaging (e.g. compression hose, custom garments, commercial kits, etc.) prior to the Baseline visit. If clinically necessary, subjects may have received other wound treatments as needed (e.g., surgical debridement, pressure off-loading, negative pressure and/or hyperbaric oxygen therapy).
* Subjects must have previously undergone venous hemodynamic correction via compression, surgical venous stripping, sclerotherapy, endovenous laser ablation, and/or endovenous radiofrequency ablation.
* Subjects must have adequate circulation to the affected extremity as demonstrated by the most recently measured ankle-brachial index (ABI) greater than or equal to 0.8 and less than or equal to 1.2 or triphasic or biphasic Doppler arterial waveforms at the ankle of the affected leg (as applicable). If subject has undergone lower extremity stenting or bypass where ABI would be considered unreliable to assess microvascular circulation, subjects must have transcutaneous oximetry (TcPO2) > 40 mmHg.
* Subjects must have VSU caused by underlying venous reflux disease with physiological reflux lasting greater than 500 milliseconds for superficial veins and 1.0 seconds for deep veins, as confirmed by most recent Doppler ultrasound venous mapping from Baseline; historical results/confirmation within the previous three years allowed.
* Subjects who agree to follow the specified precautions to avoid pregnancy as follows:

Subjects who are females of childbearing potential include any female subject who has experienced menarche and who has not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or is not postmenopausal (defined as amenorrhea for at least 12 consecutive months). For female subjects of childbearing potential, a negative urine pregnancy test is required at Screening and Baseline prior to initiating Study Product. Female subjects of childbearing potential must follow 1 of the following approaches:

* Practice actual abstinence from intercourse
* Have a partner with a vasectomy
* Have an intrauterine device
* Must use 2 different forms of highly effective contraception for the duration of the study, and for at least 48 hours after discontinuing study drug. Medically acceptable forms of effective contraception include approved hormonal contraceptives (such as birth control pills) or barrier methods (such as a condom or diaphragm).

  * Male subjects with a partner of childbearing potential must use a condom during intercourse for the duration of the study, and for 48 hours after discontinuing study drug.

    * Subjects who, in the opinion of the Investigator, are capable of communicating effectively with study personnel and are considered reliable, willing, and likely to be cooperative with protocol requirements and attend all required study visits.
    * Subjects who have the capability to answer surveys and questionnaires written in English.

Exclusion Criteria:

* Subject must not be currently receiving topical antimicrobials and ulcer must not be infected as determined by clinical assessment (e.g. odor, color, visual appearance) rather than culture.
* Ulcer must not have exposed bone, tendon, or ligament.
* Subject must not have another ulcer within 3 cm from the ulcer receiving investigational treatment.
* Female subjects who are pregnant, lactating, or planning to become pregnant during the study.
* Subjects actively receiving or received a skin graft substitutes within 30 days prior to Baseline.
* Subjects receiving oral, systemically administered, or lower extremity injectable corticosteroid therapy within 60 days prior to Baseline.

Subjects with angiographic or clinical signs of peripheral arterial disease (PAD) or congestive heart failure (CHF) with most previous echocardiogram demonstrating an ejection fraction (EF) less than 35%.

* Subjects with underlying osteomyelitis.
* Subjects with an active infection or condition that would interfere with interpretation of study assessments.
* Subjects with an HbA1c > 7.0% (Part 1 only) or HbA1c > 8.0% (Part 2 only), as collected at Screening or in the previous 120 days prior to Screening.
* Subjects with current deep vein thrombosis (DVT) (Part 2 only)
* Subjects with chronic musculoskeletal disorder or any other disease that would limit ambulation.
* Subjects with a history of alcohol abuse or illicit drug abuse within 12 months of Baseline which, in the Investigator's opinion, would make the subject inappropriate for enrollment in a clinical study.
* Subjects with any other concomitant disease with life expectancy of <12 months from Baseline
* Subjects with an unstable psychiatric condition or those not capable of understanding the objectives, nature, or consequences of the study, or who have any condition which, in the Investigator's opinion, would constitute an unacceptable risk to the subject's safety.
* Subjects who are currently receiving an investigational drug, have an investigational device in place, or who have participated in an investigational drug or device study within 90 days prior to Baseline. Participation in an observational study within 90 days prior to Baseline does not disqualify a subject from enrolling.
* Subjects who have received another regenerative therapy within 30 days prior to Baseline.
* Subjects with a Body Mass Index (BMI) > 45 (Part 2 only).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-02-26 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-10-15 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability | Baseline to Week 12
  Evaluated via patient and/or Investigator reported adverse events that occur during the study

SECONDARY OUTCOMES:
Total wound closure | Baseline to Week 12
  Total ulcer closure demonstrated by skin re-epithelization without drainage or dressing requirements at two consecutive visits > 2 weeks
Ulcer size | Baseline to Week 12
  Percent reduction of the ulcer surface area
Change in pain | Baseline to Weeks 4, 8 and 12
  Change in patient-reported index ulcer-related pain via the score from the Visual Analogue Scale (VAS)
Change in health-related quality of life | Baseline to Week 12
  SF-36, DLQI, and Wound-QOL

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - Compass Medical Research Center, Tucson, Arizona
  - Center for Clinical Research, Inc., Castro Valley, California
  - Limb Preservation Platform, Inc., Fresno, California
  - Center for Clinical Research Inc., San Francisco, California
  - Center for Clinical Research, Inc., San Francisco, California
  - Massachusetts General Hospital, Boston, Massachusetts
  - Northwell Health, Inc., New Hyde Park, New York
  - Brock Liden DPM, Circleville, Ohio
  - Salem Vamc, Salem, Virginia

IPD SHARING:
Plan to Share IPD: No